CLINICAL TRIAL: NCT06294561
Title: An Open-label, Two-cycle, Single Sequence, Self-controlled Study Evaluating Effects of Oral Itraconazole or Efavirenz on Pharmacokinetic Profiles of TGRX-326
Brief Title: TGRX-326 Pharmacokinetic Drug Interaction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen TargetRx, Inc. (Industry)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TGRX-326-1003
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Itraconazole (Experimental): healthy subjects will be given Itraconazole 200 mg orally with TGRX-326 60 mg
  Interventions: Drug: Itraconazole+TGRX-326
- Efavirenz (Experimental): healthy subjects will be given Efavirenz 600 mg orally with TGRX-326 60 mg
  Interventions: Drug: Efavirenz+TGRX-326

INTERVENTIONS:
Drug: Itraconazole+TGRX-326 — healthy subjects will be given TGRX-326 60 mg orally on Day 1, and Itraconazole 200 mg with TGRX-326 60 mg orally on day 11
  Arms: Itraconazole
Drug: Efavirenz+TGRX-326 — healthy subjects will be given TGRX-326 60 mg orally on Day 1, and Efavirenz 600 mg with TGRX-326 60 mg orally on day 20
  Arms: Efavirenz

SUMMARY:
This is a drug-drug interaction study for TGRX-326 to evaluate the effects of CYP3A inhibitor/inducer drugs on pharmacokinetic profiles of TGRX-326, an ALK inhibitor indicated for treatment of Non-small cell lung cancer.

DETAILED DESCRIPTION:
This study is designed as an open-label, single sequence, self-controlled study. The study will be conducted for 2 cycles, 10 days per cycle. Itraconazole, a CYP3A inhibitor, and Efavirenz, a CYP3A inducer, will be administrated orally with TGRX-326 to evaluate the effect of these drugs on the pharmacokinetic profiles of TGRX-326. Pharmacokinetic parameters will be evaluated as primary endpoints. Safety evaluation will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* healthy subject; male or female
* Age between 18 and 45 (inclusive)
* body mass index (BMI) between 19.0 and 26.0 (inclusive)
* agree to consent
* able to communicate with investigator well and complete the study according to study protocol

Exclusion Criteria:

* abnormal and clinically significant test results (including physical exam, laboratory tests, 12-lead ECG, chest x-ray, etc.)
* any one positive result for hepatitis-B surface antigen, Hepatitis C antibody, HIV antibody or syphilis antibody
* prolongation in QT interval
* use of substance that affects CYP3A4 enzyme activity with 30 days before screening
* use of any drug within 14 days of test article administration
* use of any investigational drug or participation of any clinical study within 3 months before screening
* vaccination within 14 days before first test article administration, or have plans to receive vaccination during the study period
* history of cardiovascular diseases
* history of mental conditions including depression, aggressive behaviours, epilepsy, etc.
* history of major surgery within 6 months before screen, or have unhealed surgical wounds.
* any clinically significant conditions that investigator believes could affect study outcomes
* history of allergic reactions, or allergic to any components to the study drugs, or have food allergy/special requirement for food that forbids the subject to follow food requirements for the study
* daily cigarette consumption of more than 5 within 3 months before screening, or cannot avoid using cigarette/tabacco products during the study
* history of alcohol abuse (more than 14 units of alcohol per week) within 3 months before screening, or alcohol breath test of > 0.0 mg/dl at screening
* history of substance abuse, or positive drug results at screening
* history of certain food intake 2 weeks before screening, and/or use of more than 8 cups of tea/coffee/grapefruit juice
* positive pregnancy test results, or pregnant/breast-feeding females
* history of unprotected sexual activities within 1 month before screening
* have plans for child bearing during study period and for 6 months after study, or disagree to take contraceptive measures during study period and for 6 months after study
* history of blood donation or blood loss within 3 months before screening, or have plans to donate blood within 1 month after the study
* any reasons that is deemed unsuitable for study participation as determined by investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Plasma Tmax | Itraconazole group: Day 1, Days 2-6, Day 11, Days 12-15 and Day 16 (or last day of dosing); Efavirenz group: Day 1, Days 2-6, Day 20, Day 21-24 and Day 25 (or last day of dosing)
  Time to maximum concentration of TGRX-326 measured in plasma
Plasma Cmax | Itraconazole group: Day 1, Days 2-6, Day 11, Days 12-15 and Day 16 (or last day of dosing); Efavirenz group: Day 1, Days 2-6, Day 20, Day 21-24 and Day 25 (or last day of dosing)
  Maximum concentration of TGRX-326 measured in plasma
Plasma AUC(0-t) | Itraconazole group: Day 1, Days 2-6, Day 11, Days 12-15 and Day 16 (or last day of dosing); Efavirenz group: Day 1, Days 2-6, Day 20, Day 21-24 and Day 25 (or last day of dosing)
  Area Under drug concentration-time curve (AUC) from time 0 to last measureable timepoint for TGRX-326 as measured in plasma
Plasma AUC(0-inf) | Itraconazole group: Day 1, Days 2-6, Day 11, Days 12-15 and Day 16 (or last day of dosing); Efavirenz group: Day 1, Days 2-6, Day 20, Day 21-24 and Day 25 (or last day of dosing)
  Area Under drug concentration-time curve from time 0 to infinity for TGRX-326 as measured in plasma
T1/2 | Itraconazole group: Day 1, Days 2-6, Day 11, Days 12-15 and Day 16 (or last day of dosing); Efavirenz group: Day 1, Days 2-6, Day 20, Day 21-24 and Day 25 (or last day of dosing)
  Plasma half-life of TGRX-326
Plasma volume of distribution (Vz/F) | Itraconazole group: Day 1, Days 2-6, Day 11, Days 12-15 and Day 16 (or last day of dosing); Efavirenz group: Day 1, Days 2-6, Day 20, Day 21-24 and Day 25 (or last day of dosing)
  Apparent volume of distribution of TGRX-326 in plasma
Plasma clearance (CL/F) | Itraconazole group: Day 1, Days 2-6, Day 11, Days 12-15 and Day 16 (or last day of dosing); Efavirenz group: Day 1, Days 2-6, Day 20, Day 21-24 and Day 25 (or last day of dosing)
  Apparent clearance of TGRX-326 in plasma

SECONDARY OUTCOMES:
Adverse events/serious adverse events | through completion of the study, an average of 1 month
  to record and analyse subjects with adverse events (AEs) and serious adverse events (SAEs)
Corrected QT Interval | At screening; Itraconazole group: Day 1, Days 2-5, Day 11, Days 12-15 and Day 16 (or last day of dosing); Efavirenz group: Day 1, Day 20 and Day 25 (or last day of dosing)
  Corrected QT Interval (QTc) as measured by 12-lead electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, MD, Principal Investigator — Nanjing Drug Tower Hospital
Locations (1):
- Nanjing Drug Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No